CLINICAL TRIAL: NCT01312324
Title: A Prospective, Phase II Trial of Induction Chemotherapy With Docetaxel/Cisplatin for Masaoka Stage III/IV Thymic Epithelial Tumors
Brief Title: Neoadjuvant Chemotherapy for Locally Advanced Thymic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Keunchil Park, Principal investigator, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-01-040
Record Dates: First submitted 2011-03-06; First posted 2011-03-10 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Locally Advanced Stage III or IV Thymic Cancer
Keywords: neoadjuvant chemotherapy; thymic cancer
MeSH Terms: conditions — Thymus Neoplasms | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- neoadjuvant chemotherapy (Experimental): 3 cycles of docetaxel/cisplatin before operation
  Interventions: Drug: neoadjuvant docetaxel/cisplatin

INTERVENTIONS:
Drug: neoadjuvant docetaxel/cisplatin — 3 cycles of docetaxel plus cisplatin docetaxel 75mg/m2 D1 cisplatin 75mg/m2 D1 every 3 weeks

SUMMARY:
We try to evaluate whether neoadjuvant docetaxel plus cisplatin can increase the complete resection rate in advanced thymic carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed thymic carcinoma
* surgically inoperable Masaoka stage III or IV
* ECOG 0-2
* at least one measurable disease

Exclusion Criteria:

* previous myocardiac infarct history within 1 year before the enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2007-02; Primary Completion 2015-07 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Complete resection rate | 4-8 weeks later after completion of neoadjuvant chemotherapy

SECONDARY OUTCOMES:
the number of patients with adverse events | from enrollment to 6 months after completion of chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea